CLINICAL TRIAL: NCT00635778
Title: An Open-Label, Dose Escalation Phase I Trial of MK-0646 Given as a One to Two Hour Every Other Week Infusion in Patients With Relapsed or Refractory Locally Advanced or Metastatic Cancers
Brief Title: A Dose-finding Study of Dalotuzumab in Subjects With Advanced Solid Tumors (MK-0646-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0646-002; MK-0646-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-14 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — dalotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- dalotuzumab 2.5/2.5 mg/kg (Experimental): Participants received a loading dose of dalotuzumab 2.5 mg/kg administered by intravenous (IV) infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 2.5 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab
- dalotuzumab 5.0/5.0 mg/kg (Experimental): Participants received a loading dose of dalotuzumab 5.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab
- dalotuzumab 10.0/5.0 mg/kg (Experimental): Participants received a loading dose of dalotuzumab 10.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab
- dalotuzumab 15.0/5.0mg/kg (Experimental): Participants received a loading dose of dalotuzumab 15.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab
- dalotuzumab 20.0/5.0 mg/kg (Experimental): Participants received a loading dose of dalotuzumab 20.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab
- dalotuzumab 15.0/10.0 mg/kg (Experimental): Participants received a loading dose of dalotuzumab 15.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 10.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab
- dalotuzumab 15.0/15.0 mg/kg (Experimental): Participants received a loading dose of dalotuzumab 15.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 15.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
  Interventions: Drug: dalotuzumab

INTERVENTIONS:
Drug: dalotuzumab — Administered as an IV infusion over one to two hours
  Other Names: MK-0646

SUMMARY:
The study determined the recommended Phase 2 loading and maintenance doses and dose schedules for administering dalotuzumab using dose-limiting toxicities (DLTs) observed during the entire treatment period (Up to 18 months). The primary hypothesis of the study was that administration of dalotuzumab as an every other week infusion in participants with relapsed or refractory locally advanced or metastatic cancers associated with a high frequency of insulin-like growth factor receptor type 1(IGF-1R) overexpression will be generally safe and well tolerated to permit further study and achieve a constant clearance and a minimum trough concentration of 3 µg/mL.

DETAILED DESCRIPTION:
The study consisted of 3 parts. In Part 1 the loading dose was escalated while the maintenance dose was kept constant. In Part 2 the loading dose was kept constant while the maintenance dose was escalated. In Part 3 the recommended phase 2 loading and maintenance doses and schedule were administered to an expanded cohort to explore safety and efficacy of dalotuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with advanced solid tumors who have failed to respond to standard therapy, ages 18 years and older, with adequate organ function

Exclusion Criteria:

* Participant is using growth hormones or growth hormone inhibitors
* Participant is known to be allergic to components of the drug or similar drugs (e.g. monoclonal antibodies such as rituximab or biological therapies such as immunoglobulin G
* Participant has had chemotherapy, radiotherapy, or biological therapy within 4-6 weeks of entering the study or has not recovered from previous therapy
* Participant is taking part in or has taken part in a study of an investigational compound or device within 30 days of their first dose of study drug
* Participant has an active Central Nervous System metastases and/or carcinomatous meningitis. However, a participant who has completed a course of therapy and is clinically stable may be able to participate
* Participant is pregnant or breastfeeding
* Participant is human immunodeficiency virus (HIV) positive
* Participant has a history of Hepatitis B or C
* Participant has symptomatic ascites or pleural effusion. However, if the participant has received treatment and is stable, they may be able to participate
* Female participant plans to become pregnant or a male participant who plans to impregnate their partner during the time the study is ongoing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08-07 (Actual); Primary Completion 2008-11-05 (Actual); Study Completion 2008-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with metastatic or locally advanced solid tumors, associated with insulin-like growth factor receptor type 1 (IGF-1R) protein expression, that have failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist. Other inclusion/exclusion criteria applied.
Groups:
- Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg: Participants received a loading dose of dalotuzumab 2.5 mg/kg administered by intravenous (IV) infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 2.5 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg: Participants received a loading dose of dalotuzumab 5.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg: Participants received a loading dose of dalotuzumab 10.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg: Participants received a loading dose of dalotuzumab 15.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg: Participants received a loading dose of dalotuzumab 20.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 5.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg: Participants received a loading dose of dalotuzumab 15.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 10.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg: Participants received a loading dose of dalotuzumab 15.0 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 15.0 mg/kg administered by IV infusion every two weeks for up to 18 months.
Period: Overall Study
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg
Started | 1 | 3 | 3 | 8 | 8 | 21 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 3 | 8 | 8 | 21 | 6
Not completed — Adverse Event | 1 | 0 | 0 | 3 | 3 | 6 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Progressive disease | 0 | 3 | 3 | 4 | 5 | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg: Participants received a loading dose of dalotuzumab 2.5 mg/kg administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab 2.5 mg/kg administered by IV infusion every two weeks for up to 18 months.
- Total: Total of all reporting groups
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg | Total
Number analyzed (Participants) | 1 | 3 | 3 | 8 | 8 | 21 | 6 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (NA) — Not calculated for only 1 participant | 74.3 (9.9) | 60.3 (8.6) | 71.3 (6.5) | 59.1 (7.6) | 58.1 (11.8) | 53.7 (21.2) | 61.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 1 | 10 | 2 | 17
  Male | 1 | 2 | 1 | 7 | 7 | 11 | 4 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of participants is presented. Population: All enrolled participants.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    White | 1 | 3 | 2 | 6 | 4 | 17 | 5 | 38
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 7
Number of Prior Chemotherapy Regimens [Mean (Standard Deviation); unit: Regimens] | 3.0 (NA) — Not calculated on only 1 participant | 2.7 (0.6) | 3.0 (0.0) | 3.0 (0.0) | 3.0 (0.0) | 2.9 (0.3) | 2.5 (0.8) | 2.9 (0.4)
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all self-care but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any self-care, totally confined to bed or chair or Grade 5: Dead. Population: All enrolled participants
  Participants
    ECOG PS = 0 | 0 | 1 | 1 | 1 | 3 | 10 | 4 | 20
    ECOG PS = 1 | 0 | 2 | 2 | 6 | 5 | 10 | 1 | 26
    ECOG PS = 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Serum Concentration of Dalotuzumab at 336 Hours (C336) After the First Maintenance Dose
Description: Blood samples were obtained for analysis of steady-state serum concentration of dalotuzumab at 336 hours (C336) after the first maintenance dose of dalotuzumab. The C336 of dalotuzumab after intravenous administration is presented.
Time Frame: 2 weeks post first maintenance dose of study drug (3 weeks post loading dose of study drug)
Population: All participants who received dalotuzumab and had blood samples drawn for pharmacokinetic (PK) analyses.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 6 | 8 | 19 | 5
μg/mL | 4.78 (NA) — Not calculated on only 1 participant | 7.48 (8.50) | 54.57 (24.64) | 33.00 (24.90) | 25.95 (26.22) | 24.39 (27.63) | 86.73 (44.56)

2. Primary Outcome: Number of Participants Who Experience One or More Dose- Limiting Toxicities (DLTs)
Description: Dose-limiting toxicities (DLT) were assessed and graded using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE). A DLT was defined as the occurrence of any of the following events, that were judged by the study investigator, to be related to the study medication: Grade 4 neutropenia; Grade 3 neutropenia with fever >38.5 degrees Celsius; Grade 4 thrombocytopenia; Grade 3 or Grade 4 non-hematologic toxicity (except alopecia and inadequately treated diarrhea, nausea, and vomiting, and hyperglycemia lasting less than 5 days; and Grade 3 or greater hyperglycemia lasting for more than 5 days in spite of optimal medical management.
Time Frame: The entire treatment period (Up to 18 months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg
Number analyzed (Participants) | 1 | 3 | 3 | 8 | 8 | 21 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants Who Experienced a Complete Response (CR) or Partial Response (PR)
Description: Complete Response (disappearance of all target lesions) or Partial Response (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) using Response Criteria in Solid Tumors (RECIST). Tumor response was assessed prior to first dose and every 8 weeks beginning pre-dose of Week 9 for up to 18 months. The best response out of all measurements for each participant was used for determining CR and PR.
Time Frame: Up to 18 months post first dose of study drug
Population: All participants who received at least one dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg
Number analyzed (Participants) | 1 | 3 | 3 | 8 | 8 | 21 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Serum Insulin-like Growth Factor Receptor Type 1 (IGF-1R) Protein Level at Week 1
Description: IGF-1R expression was measured in pre- and post-dose biopsy samples using immunohistochemistry (IHC) and enzyme-linked immunosorbent assay (ELISA) assays. Results were expressed as a percent change from baseline in IG1-FR expression for participants pooled across all dose arms in the study and calculated by study week. A post-dose decrease in IGF-1R expression was an indication of target engagement by dalotuzumab. A larger percent change correlated with a greater target engagement.
Time Frame: Baseline and Week 1
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 1.
Measure: Median (Full Range); unit: Percent change
Groups:
- Pooled Participants Who Received Dalotuzumab: Participants were pooled from all dose arms in the study. Participants received a loading dose of dalotuzumab administered by IV infusion. Two weeks following completion of the loading dose, participants received a maintenance dose of dalotuzumab administered by IV infusion every two weeks for up to 18 months.
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 41
Percent change | 118.56 [-61.54 to 377.08]

5. Secondary Outcome: Number of Participants With a Positive Human-anti-humanized-antibody (HAHA) Titer
Description: The formation of HAHAs may block efficacy by prematurely clearing dalotuzumab and limit the possibility of future dalotuzumab therapy. Blood samples for the measurement of serum levels of HAHAs were obtained prior to treatment with dalotuzumab, and pre-dose Week 3, Week 5, pre-dose every 8 subsequent weeks, and end of treatment (post-study: 4 weeks after last dose of study drug). Positive HAHA status for a participant is defined as testing positive on both the screening and immunodepletion assays at one or more visits.
Time Frame: Prior to second and subsequent doses of study drug (Up to 1 year post-first dose)
Population: All participants who received one dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg
Number analyzed (Participants) | 1 | 3 | 3 | 8 | 8 | 21 | 6
Participants | 0 | 0 | 0 | 2 | 1 | 1 | 0

6. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 5
Description: as for outcome 4
Time Frame: Baseline and Week 5
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 5
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 25
Percent change | 150.94 [-49.35 to 421.84]

7. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 9
Description: as for outcome 4
Time Frame: Baseline and Week 9
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 9
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 6
Percent change | 150.69 [55.00 to 246.51]

8. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 13
Description: as for outcome 4
Time Frame: Baseline and Week 13
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 13
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 4
Percent change | 138.11 [128.42 to 164.29]

9. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 17
Description: as for outcome 4
Time Frame: Baseline and Week 17
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 17
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 3
Percent change | 140.72 [120.00 to 198.05]

10. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 21
Description: as for outcome 4
Time Frame: Baseline and Week 21
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 21
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 3
Percent change | 150.00 [102.40 to 161.05]

11. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 25
Description: as for outcome 4
Time Frame: Baseline and Week 25
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 25
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 3
Percent change | 157.49 [114.74 to 170.78]

12. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 29
Description: as for outcome 4
Time Frame: Baseline and Week 29
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 29
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 2
Percent change | 174.95 [172.63 to 177.27]

13. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 33
Description: as for outcome 4
Time Frame: Baseline and Week 33
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 33
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 1
Percent change | 158.95 [NA to NA] — Not calculated on only 1 participant

14. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 37
Description: as for outcome 4
Time Frame: Baseline and Week 37
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 37
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 1
Percent change | 186.32 [NA to NA] — Not calculated on only 1 participant

15. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 41
Description: as for outcome 4
Time Frame: Baseline and Week 41
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 41
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 1
Percent change | 173.68 [NA to NA] — Not calculated on only 1 participant

16. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 45
Description: as for outcome 4
Time Frame: Baseline and Week 45
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 45
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 1
Percent change | 140.00 [NA to NA] — Not calculated on only 1 participant

17. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 49
Description: as for outcome 4
Time Frame: Baseline and Week 49
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 49
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 1
Percent change | 137.89 [NA to NA] — Not calculated on only 1 participant

18. Secondary Outcome: Percent Change From Baseline in Serum IGF-1R Protein Level at Week 53
Description: as for outcome 4
Time Frame: Baseline and Week 53
Population: All participants who took at least one dose of study drug and had available IGF-1R protein data for Baseline and Week 53
Measure: Median (Full Range); unit: Percent change
Arm/Group | Pooled Participants Who Received Dalotuzumab
Number analyzed (Participants) | 1
Percent change | 198.99 [NA to NA] — Not calculated on only 1 participant

ADVERSE EVENTS:
Time Frame: Up to 19 months (up to 18 months of treatment with study drug plus 1 month of follow-up)
Description: The safety population consisted of all participants who received at least one dose of study drug.
Arm/Group | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/3 | 0/3 | 1/8 | 1/8 | 1/21 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/3 | 2/3 | 5/8 | 6/8 | 9/21 | 3/6
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 8/8 | 8/8 | 21/21 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg (N=1) | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=3) | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=3) | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=8) | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=8) | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg (N=21) | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 2.5 mg/kg / Dalotuzumab 2.5 mg/kg (N=1) | Dalotuzumab 5.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=3) | Dalotuzumab 10.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=3) | Dalotuzumab 15.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=8) | Dalotuzumab 20.0 mg/kg / Dalotuzumab 5.0 mg/kg (N=8) | Dalotuzumab 15.0 mg/kg / Dalotuzumab 10.0 mg/kg (N=21) | Dalotuzumab 15.0 mg/kg / Dalotuzumab 15.0 mg/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 6 (6) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myodesopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (3) | 1 (1) | 2 (2) | 10 (10) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 7 (10) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (7) | 3 (3) | 12 (12) | 4 (4)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Portal vein occlusion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (5) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (6) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haemoglobin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (5) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 4 (6) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asterixis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.